CLINICAL TRIAL: NCT03985488
Title: Prospective Registry of Radiation Exposure Measurement in Procedures Utilizing Fluoroscopy
Brief Title: Radiation Exposure Assessment in Fluoroscopy
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1434665
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Fluoroscopy; Adverse Effect; Radiation Exposure
Keywords: endoscopy; fluoroscopy; radiation exposure
MeSH Terms: interventions — Radiation Exposure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eview Fluoroscopy Machine: The Eview Fluoroscopy Machine is the standard of care fluoro machine used in endoscopy.
  Interventions: Radiation: Radiation exposure
- Fluoroshield Device: The FluoroShield technology (Omega Medical Imaging) has been developed in an effort to further reduce the degree of radiation exposure to patients and provides. This technology is an additional component that can be fitted to the preexisting Eview fluoroscopy machines, in order to further filter radiation that has passed through the pre-existing machine.
  Interventions: Radiation: Radiation exposure

INTERVENTIONS:
Radiation: Radiation exposure — Radiation exposure via Eview Fluoroscopy machine.

SUMMARY:
There has been increasing awareness regarding the risk of radiation exposure to patients and providers when performing procedures requiring fluoroscopic guidance.

DETAILED DESCRIPTION:
Fluoroscopy guidance is routinely used in many endoscopic procedures per standard-of-care practice and there is increasing effort to minimize the degree of radiation exposure to patients and providers during fluoroscopy usage. The current fluoroscopy machine used per standard-of-care practice at the Center for Interventional Endoscopy is the Eview machine (Omega Medical Imaging, Orlando, FL, USA). Recently, CA-100S technology (FluoroShield, Omega Medical Imaging) has been developed in an effort to further reduce the degree of radiation exposure to patients and provides. This technology is an additional component that can be fitted to the preexisting Eview fluoroscopy machine, in order to further filter radiation that has passed through the pre-existing machine. The investigators will be performing this study to determine the degree of radiation exposure to patients and providers when using the Eview fluoroscopy machine, with and without the FluoroShield radiation exposure reduction system.

There has been increasing awareness regarding the risk of radiation exposure to patients and providers when performing procedures requiring fluoroscopic guidance. In a prior study, the Eview machine, which is currently used for fluoroscopy guidance at the Center for Interventional Endoscopy, was shown to decrease, but not completely eliminate, radiation exposure when compared to C-arm type of fluoroscopy machines (GE Healthcare, Wauwatosa, WI, USA). Recently, the FluoroShield technology (Omega Medical Imaging) has been developed in an effort to further reduce the degree of radiation exposure to patients and provides. This technology is an additional component that can be fitted to the preexisting Eview fluoroscopy machines, in order to further filter radiation that has passed through the pre-existing machine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Having an endoscopy with fluoroscopy

Exclusion Criteria:

* Less than 18 years of age
* Not having an endoscopy with fluoroscopy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is any patient that is having an endoscopy with fluoroscopy at the site.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Degree of exposure measured by Dap meter and cumulative air KERMA | 1 day
  Measurement of the degree of radiation exposure to patients and providers when performing endoscopic procedures with fluoroscopy guidance, with and without the FluroShield radiation exposure reduction system will be measured. The data will be collected in microgray per meter squared (Dap meter) and milligray (cumulative air KERMA).

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Bang JY, Hough M, Hawes RH, Varadarajulu S. Use of Artificial Intelligence to Reduce Radiation Exposure at Fluoroscopy-Guided Endoscopic Procedures. Am J Gastroenterol. 2020 Apr;115(4):555-561. doi: 10.14309/ajg.0000000000000565. PMID 32195731